CLINICAL TRIAL: NCT01446536
Title: Decreased Readmissions and Improved Quality of Care With Use of Inexpensive Checklist in Heart Failure
Brief Title: Effect of Quality Improvement Tools in Congestive Heart Failure (CHF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph Mercy Oakland Hospital (Other)
Responsible Party: Principal Investigator, Abhijeet Basoor, Cardiology Fellow, St. Joseph Mercy Oakland Hospital
Masking: Single
Other Study IDs: 11-09-02
Record Dates: First submitted 2011-09-30; First posted 2011-10-05 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Congestive Heart Failure
Keywords: Quality; Improvement
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Control group (No Intervention): This arm which was control group, was randomly selected among patients with acute decompensated heart failure in whom the checklist was not used. This group was managed as per the standard guidelines.
- Checklist (intervention) cohort (Active Comparator): checklist was used in this group arbitrarily by their treating physician
  Interventions: Other: Checklist cohort

INTERVENTIONS:
Other: Checklist cohort — CHF discharge checklist was used arbitrarily by their treating physicians in addition to the standard therapy
  Arms: Checklist (intervention) cohort

SUMMARY:
Hypothesis: Quality Improvement tools like "Heart Failure Discharge Checklist" which emphasizes on proper education to patients, ensure appropriate dose titration and counselling improve outcome in congestive heart failure (CHF).

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to SJMO with principal diagnosis of acute decompensated heart failure

Exclusion Criteria:

* Age less than 18 years
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2008-08; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Readmissions | 6 months
  Readmission to the hospital for CHF within 6 months of discharge
Dose titration | patients were followed during the time of hospital stay, average of 5 days
  up titration of medications including Beta blocer, ACE inhibitor or ARB was assessed during the hospital stay

SECONDARY OUTCOMES:
Medications prescribed | patients were followed during their hospital stay from admission to discharge, on an average of 5 days
  during the hospital stay and at discharge this outcome is measured/assessed

CONTACTS AND LOCATIONS:
Overall Officials: Abhijeet Basoor, MD, Principal Investigator — St. Joseph Mercy Oakland Hospital
Locations (1):
- St. Joseph Mercy Oakland Hospital, Pontiac, Michigan, United States